CLINICAL TRIAL: NCT06009757
Title: Safety and Efficacy of the GUIDEX® Versus Launcher™ Guiding Catheter in Adults' Patients With Coronary Artery Disease (CAD) Requiring Percutaneous Coronary Intervention (PCI): a Non-inferiority and Randomized, Clinical Trial.
Brief Title: GUIDEX® Versus Launcher™ Guiding Catheter in Percutaneous Coronary Intervention (PCI) (GUIDEX_FR)
Acronym: GUIDEX®_FR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Demax Medical Technology Co., Ltd (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Organization: DemaxGroup (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLI-00910
Record Dates: First submitted 2023-07-28; First posted 2023-08-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Guiding catheter
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Thus the aim of this non-inferiority study is to compare the efficacy and safety for patients with coronary artery disease during a percutaneous coronary intervention between Guidex® Guiding catheter (DEMAX) and Launcher™ coronary guide catheters (Medtronic).
Who Masked: Participant
Masking Description: The study is single-blind. The patient does not know which guidance catheter will be used.
  Due to the nature of the intervention (different form of guiding catheter), staff may not be blind to the allocation, but they are strongly encouraged not to disclose the participant's allocation status during follow-up assessments. The sponsor's team will not know what type of treatment the patient's number corresponds to. Under no circumstances will they have access to the list of matches between the patient number and the allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Coronary Intervention with Guiding Catheter GUIDEX (Experimental): Patients with coronary artery disease during a percutaneous coronary intervention will be treated with one of the guiding catheter
  Interventions: Device: GUIDEX® guiding catheter
- Percutaneous Coronary Intervention with Guiding Catheter Medtronics (Experimental): Patients with coronary artery disease during a percutaneous coronary intervention will be treated with one of the guiding catheter
  Interventions: Device: Launcher™ coronary guide catheter

INTERVENTIONS:
Device: GUIDEX® guiding catheter — The main steps of the procedure Percutaneous Coronary Intervention are :
  * The patient should prepare for angioplasty using standard techniques. Appropriate anticoagulation and vasodilation therapy should be administered.
  * The Guiding Catheter must be introduced into the vascular system by cut-down or percutaneous techniques.
  * The guiding catheter will be introduce over a previously placed standard angiographic wire. It will be aspirate and flush after the removal of the angiographic wire following established angiographic technique.
  * The catheter should should address the selected vascular site
  * The guiding catheter will be removing. The procedure is performed in a healthcare facility, in an operating room under fluoroscopic monitoring. The users are trained practiticoners for PCI.
  Arms: Percutaneous Coronary Intervention with Guiding Catheter GUIDEX
Device: Launcher™ coronary guide catheter — The main steps of the procedure Percutaneous Coronary Intervention are :
  * The patient should prepare for angioplasty using standard techniques. Appropriate anticoagulation and vasodilation therapy should be administered.
  * The Guiding Catheter must be introduced into the vascular system by cut-down or percutaneous techniques.
  * The guiding catheter will be introduce over a previously placed standard angiographic wire. It will be aspirate and flush after the removal of the angiographic wire following established angiographic technique.
  * The catheter should should address the selected vascular site
  * The guiding catheter will be removing. The procedure is performed in a healthcare facility, in an operating room under fluoroscopic monitoring. The users are trained practiticoners for PCI.
  Arms: Percutaneous Coronary Intervention with Guiding Catheter Medtronics

SUMMARY:
The goal of this clinical trial is to compare two guiding catheters in patients with coronary artery disease during a percutaneous coronary intervention between Guidex® Guiding catheter (DEMAX) and Launcher™ coronary guide catheters (Medtronic). The main question[s] it aims to answer are:

* Aren't the safety of medical devices inferior to each other?
* Aren't the efficacyof medical devices inferior to each other? Participants will be randomized (1:1) and have a percutaneous coronary interventionwith one of the two guiding catheters.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the most common cause of death in the European region. In line with the Global Burden of Disease (GBD) estimates from 2001, 43% of all Cardio Vascular Disease (CVD) deaths are related to coronary artery disease (CAD).

Treatment of CAD is always based on medication, which may also be supplemented by invasive procedures. The most significant historical advances in the treatment of coronary artery disease were the development of coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI).

An essential element in the success of an angioplasty and in shortening the procedure, the guiding catheter is not simply a support. While, it's primary role is designed to provide a pathway through which balloon dilation catheter, guide wire or other devices are introduced, it can also contribute to significant semantic information since it is the first tool to appear in the field of view. A variety of guiding catheter references are available on the market.

Guiding catheters of various sizes and shapes are selected based on vessel anatomy, lesion characteristics, vascular access and procedural complexity.

The GUIDEX® device is a guiding catheter designed to be used in percutaneous coronary intervention. GUIDEX® device is on the Chinese market since September 2015 (certificate renewal in 2020) and is presented for CE marking according to MDR 2017/745.

The aim of the study is to assess the essential requirements for CE marking of Guidex®: the efficacy and safety of the device. Thus the aim of this non-inferiority study is to compare the efficacy and safety for patients with coronary artery disease during a percutaneous coronary intervention between Guidex® Guiding catheter (DEMAX) and Launcher™ coronary guide catheters (Medtronic).

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be at least 18 years old.
* Patients with significant coronary artery disease who qualify for PCI (according to ACC/AHA/SCAI 2021 guidelines, including that the patient has received medical therapy with exercise and dietary recommendations before or at the same time as the PCI decision and that the clinical decision depends on the cardiology team) and who can be treated with a radial and femoral approach
* Patients scheduled for for Percutaneous Coronary Intervention and must remain overnight for observation
* The target vessel must have a TIMI flow 3 at baseline
* Palpable radial or fermoral artery
* Patients covered by the social security system

Exclusion Criteria:

* Concomitant use of Atherectomy, specialty balloon (intravascular lithotripsy), or investigational coronary devices (intravascular ultrasound, or optical coherence tomography)
* Active bleeding or significant increased risk of bleeding, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy.
* Prior PCI procedure within the last 30 days of the index procedure
* Current platelet count <100 x 10^9cells/L or Hgb <10 g/dL.
* Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
* Target vessel < 2.4 mm in diameter
* Target lesion > 32 mm in length
* Patient has allergy to imaging contrast media for which they cannot be pre-medicated
* Patients with hypersensitivity or contraindication to antiplatelet treatment
* Patient unable to stop his or her daily oral medication includes metformin treatment during 48 hours.
* Unstable patient: myocardial infarction, cardiogenic shock or with troponin above the upper limit of the normal laboratory value in the 24 hours prior to the procedure OR with elevated troponin and abnormal concomitant CK (non-exhaustive list).
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Patients who cannot read or write french;
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the frequency of in-hospital major adverse cardiac events (MACE) | Baseline until the end of the procedure
  Analyze the frequency of major adverse cardiac events (MACE) during the procedure. MACE was defined as the following:
  * Cardiac death
  * Myocardial infarction - defined as a CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave
  * TVR - defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure

SECONDARY OUTCOMES:
Percentage of subjects achieving angiographic with sucess | Baseline until End of the procedure
  The percentage of subjects achieving angiographic success were defined as success in facilating delivery of the balloon dilation catheter, guidewire or other devices introduced in the coronary arteries, using the medical devices with <50% residual stenosis without serious angiographic complications. Serious angiographic complications defined as severe dissection (Type D to F - To confirm ), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
Frequency of in-hospital major adverse cardiac events (MACE). MACE was defined as the following: a composite of cardiac death, myocardial infarction, and target lesion revascularization. | Baseline until discharge from the hospital (Day 2)
  Analyze the frequency of in-hospital major adverse cardiac events (MACE). MACE was defined as the following:
  * Cardiac death
  * Myocardial infarction - defined as a CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave
  * TVR - defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Incidence of complication and adverse event rates | [Time frame; to the baseline up to 30 days after the procedure)
  Incidence of adverse event during 1 month after the PCI (in particular related to the potential adverse event at the puncture site).
Time used for the procedure (in minutes) . | Baseline until end of the procedure (Day 1)
  Time (in minutes) between the start of the procedure until the end of the procedure
Frequency of access-site-related complications. | Baseline until End of the procedure
  The frequency of access-site related complications is defined as bleeding, pseudoaneurysm, arteriovenous fistula, and occlusion of the radial artery), which were considered to be major if they were associated with a vascular repair or a blood transfusion.
Frequency of access-site-related complications | Baseline until end of the procedure (Day 1)
  Analyse the level of angulation of the coronary artery (in degrees) during the PCI
Assessed as Fluoroscopy time (in sec) | Baseline until end of the procedure (Day 1)
  Assessed as fluoroscopy time (in sec) during the PCI

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No
Nothing